CLINICAL TRIAL: NCT04323839
Title: PRIORITY (Pregnancy Coronavirus Outcomes Registry)
Brief Title: COVID-19 PRIORITY (Pregnancy CoRonavIrus Outcomes RegIsTrY)
Acronym: PRIORITY
Status: Completed | Type: Observational
Sponsor: University of California, San Francisco (Other)
Collaborators: University of California, Los Angeles (Other)
Responsible Party: Sponsor
Other Study IDs: 20-30410
Record Dates: First submitted 2020-03-24; First posted 2020-03-27 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Pregnancy; Coronavirus; COVID-19
MeSH Terms: conditions — Coronavirus Infections; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pregnant Women: Women who are currently pregnant and are suspected or diagnosed COVID-19 positive.
  Interventions: Other: Pregnant women under investigation for Coronavirus or diagnosed with COVID-19
- Post-partum women: Women who have been pregnant in the past 6 weeks and are suspected or diagnosed COVID-19 positive.
  Interventions: Other: Postpartum women under investigation for Coronavirus or diagnosed with COVID-19

INTERVENTIONS:
Other: Pregnant women under investigation for Coronavirus or diagnosed with COVID-19 — This is an observational study with no intervention
  Groups: Pregnant Women
Other: Postpartum women under investigation for Coronavirus or diagnosed with COVID-19 — This is an observational study with no intervention
  Groups: Post-partum women

SUMMARY:
PRIORITY (Pregnancy CoRonavIrus Outcomes RegIsTrY) is a prospective cohort study of pregnant and recently pregnant women who are: either patients under investigation for COVID-19 or a confirmed case of COVID-19. Data from PRIORITY will be used to evaluate the impact of COVID-19 on the clinical course and pregnancy outcomes of pregnant women and women within 6 weeks of pregnancy.

DETAILED DESCRIPTION:
The investigators will recruit women age 13 or older under investigation for COVID-19 or with confirmed COVID-19 at any clinical state across the United States. Eligible participants will be identified through voluntary physician referrals.

When an eligible patient is referred to the PRIORITY Coordinating Center at UCSF, a UCSF study coordinator will follow-up by phone with the patient and consent verbally. The participant will be asked to complete an approval to release medical information. The investigators will use patient questionnaires to assess symptoms, maternal clinical course, pregnancy outcomes, and neonatal outcomes from initial investigation of COVID-19 to 12 months. The investigators will also obtain all medical records for the participant to data abstract key clinical and pregnancy outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Pregnant women or women who have been pregnant within the last 6 weeks
2. Able to give informed consent
3. Diagnosed with COVID-19; or being evaluated for COVID-19 ("patient under investigation") since January 1, 2020

Exclusion Criteria:

1. <13 years of age.

Min Age: 13 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Persons assigned gender female at birth.
Study Population: Pregnant women or women who have been pregnant in the last 6 weeks and are under investigation for COVID-19 or who have tested positive for COVID-19.
Sampling Method: Non-Probability Sample
Enrollment: 1333 (Actual)
Dates: Start 2020-03-20 (Actual); Primary Completion 2022-04-26 (Actual); Study Completion 2022-04-26 (Actual)

PRIMARY OUTCOMES:
Clinical presentation | Baseline to 12 months
  presenting symptoms and testing
Disease prognosis outcomes | Baseline to 12 months
  Clinical outcomes with resolution of illness
Pregnancy outcomes | Baseline to 12 months
  Pregnancy outcomes among women infected with COVID-19
Obstetric outcomes | Baseline to 12 months
  Obstetric outcomes among women infected with COVID-19
Neonatal outcomes | Baseline to 12 months
  Neonatal outcomes among infants born to women with COVID-19
Modes of transmission of COVID-19 | Baseline to 12 months
  Transmission of COVID-19 from mother to infant

CONTACTS AND LOCATIONS:
Overall Officials: Vanessa Jacoby, MD, MAS, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Afshar Y, Gaw SL, Flaherman VJ, Chambers BD, Krakow D, Berghella V, Shamshirsaz AA, Boatin AA, Aldrovandi G, Greiner A, Riley L, Boscardin WJ, Jamieson DJ, Jacoby VL; Pregnancy CoRonavIrus Outcomes RegIsTrY (PRIORITY) Study. Clinical Presentation of Coronavirus Disease 2019 (COVID-19) in Pregnant and Recently Pregnant People. Obstet Gynecol. 2020 Dec;136(6):1117-1125. doi: 10.1097/AOG.0000000000004178. PMID 33027186